CLINICAL TRIAL: NCT05483504
Title: Phase I Clinical Study to Evaluate the Tolerability, Safety, Pharmacokinetics and Immunogenicity of F61 Injection After a Single Dose in Healthy Chinese Subjects
Brief Title: Clinical Study of F61 Injection in Healthy Chinese Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wuhan Institute of Biological Products Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F61-01
Record Dates: First submitted 2022-07-27; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- F61 injection (Active Comparator): F61 injection, specification: 150 mg/5ml/bottle, batch number: 202202002-1, produced by Wuhan Institute of Biological Products Co., Ltd.
  Validity period: 24 months; Storage conditions: 2~8°C, protected from light and sealed.
  Interventions: Drug: F61 injection
- F61 placebo (Placebo Comparator): F61 placebo, specification: 5 ml/bottle, produced by Wuhan Institute of Biological Products Co., Ltd.
  Validity period: 24 months; Storage conditions: 2~8°C, protected from light and sealed.
  Interventions: Drug: F61 Placebo

INTERVENTIONS:
Drug: F61 injection — Colorless or slightly yellow liquid, may be slightly opalescent
  Arms: F61 injection
Drug: F61 Placebo — Colorless or slightly yellow liquid, may be slightly opalescent
  Arms: F61 placebo

SUMMARY:
Main purpose： To evaluate the safety and tolerability of single-dose ascending intravenous infusion of F61 in healthy subjects.

Secondary purpose： To evaluate the pharmacokinetic profile and immunogenicity of F61 administered by single ascending intravenous infusion in healthy subjects.

Research design： This study is a single-center, randomized, double-blind, placebo-controlled, single-dose escalating first-in-human Phase I trial to evaluate the tolerability, safety, and pharmacokinetics of F61 injection (F61) in healthy subjects Characteristics and Immunogenicity.

Test drug： F61 injection, specification: 150 mg/5ml/bottle, batch number: 202202002-1, produced by Wuhan Institute of Biological Products Co., Ltd.

Validity period: 24 months; Storage conditions: 2~8°C, protected from light and sealed.

Control drug： F61 placebo, specification: 5 ml/bottle, produced by Wuhan Institute of Biological Products Co., Ltd.

Validity period: 24 months; Storage conditions: 2~8°C, protected from light and sealed.

No statistical assumptions

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects aged 18-45 years (including the cut-off value);
2. The weight of male subjects is not less than 50.0 kg, and the weight of female subjects is not less than 45.0 kg, and the upper limit of acceptable weight is 80.0 kg. Body mass index (BMI) = body weight (kg)/height 2 (m2), with a BMI in the range of 18.0-28.0 kg/m2 (including critical values);
3. Physical examination, vital signs, laboratory examinations and other auxiliary examinations (frontal and lateral chest X-ray, abdominal B-ultrasound, 12-lead electrocardiogram, etc.) are normal or have no clinical significance;
4. Subjects (including partners) have no plans to become pregnant and voluntarily take effective contraceptive measures from the time of signing informed consent to the administration of the study drug within 6 months; The subjects can understand the research content and voluntarily sign the informed consent; at the same time, they can complete the research according to the requirements of the protocol.

Exclusion Criteria:

1. Those who have been diagnosed with new coronavirus pneumonia cases or suspected cases, who have had contact with confirmed or suspected cases of new coronavirus within 14 days before signing the informed consent form, or who have traveled abroad in areas with high epidemic incidence; or who have been infected with new coronavirus or carrier;
2. Patients with clinically significant abnormalities in the cardiovascular system, respiratory system, digestive system, endocrine system (diabetes), nervous/mental system, blood and lymphatic system (immune system deficiency), and skeletal muscle system confirmed by researchers ;
3. Positive results of any of the combined detection of hepatitis B surface antigen [HBsAg], hepatitis C virus antibody [Anti-HCV], human immunodeficiency virus [HIV] antigen and antibody, and Treponema pallidum specific antibody [TP-Ab];
4. Those who are known to have a history of allergies to the test drugs or excipients, or have allergies;
5. Those who have a history of vaccination within 3 months before screening, or those who have any vaccination plan during the clinical trial;
6. Those who received chemotherapy, radiotherapy, immunosuppressive therapy or high-dose corticosteroid therapy within 5 years before screening;
7. Have taken any over-the-counter, prescription, traditional Chinese medicine or vitamin within 1 month before screening;
8. Those who plan to operate during the trial;
9. Those who have a history of drug abuse or a positive urine drug screening test within 12 months before screening;
10. Regular drinkers within 6 months prior to screening, i.e. drinking more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of spirits with 40% alcohol content or 150 mL of wine), or who cannot be guaranteed to give up during the trial Alcoholic drinkers, or those with a positive breath test for alcohol;
11. Those who smoked ≥5 cigarettes per day in the 3 months before screening or those who cannot guarantee to give up smoking during the trial;
12. Those who have participated in clinical trials of other drugs within 3 months before screening (the last visit of the last trial is the start time);
13. Those who donated blood or lost more than 450 mL of blood within 3 months before screening;
14. Those who received ≥2 units of blood products within 3 months before screening;
15. Those who use tobacco, alcohol or caffeinated beverages, or strenuous exercise, or other factors that affect drug absorption, distribution, metabolism, and excretion within 24 hours before the test administration and during the test;
16. Those who plan to participate in vigorous exercise during the test, including contact sports or collision sports;
17. Women who are pregnant or breastfeeding, or those who have a positive pregnancy test result before the test; those who cannot take a medically approved non-drug contraceptive measure during the test according to the requirements of the investigator, or those who have Sperm/egg donation planners (from signing the informed consent form to within 6 months after the end of the trial);
18. Difficulty in venous blood collection or fainting of needles; The investigators think that they are not suitable to participate in this clinical trial (such as infirmity, poor compliance, etc.).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
adverse events | 105 days
  Descriptive statistics of the number of adverse events
adverse reactions | 105 days
  Descriptive statistics of the number of adverse reactions

IPD SHARING:
Plan to Share IPD: No